CLINICAL TRIAL: NCT02148081
Title: Functional Recovery in Critically Ill Children - a Longitudinal Multicentre, Mixed-Methods Study
Brief Title: Functional Recovery in Critically Ill Children, the Wee-Cover Multicentre Study
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: McMaster Children's Hospital (Other); London Health Sciences Centre (Other); Canadian Critical Care Trials Group (Other)
Responsible Party: Sponsor
Other Study IDs: 14-214
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Critical Illness
Keywords: pediatrics, critical illness, recovery, function, health
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill children

SUMMARY:
When children suffer from a critical-illness, the investigators focus on resuscitating and saving lives. Once these children leave the pediatric intensive care unit, very little is known about what happens to them - how long it takes for them to recover, how families cope, and what factors that impede their recovery. The specific objective of this research project is to evaluate how children and their families recover after a critical illness.

Research Hypotheses: Following a critical illness in children, 1) the rate and degree of health and functional recovery is influenced by the following factors: age, pre-admission co-morbid status, critical illness severity, discharge functional status, and time to initiating acute rehabilitation; 2) functional recovery is influenced by caregiver burden and health-related quality-of-life (HRQoL).

DETAILED DESCRIPTION:
The Specific Objective of this study is to evaluate the trajectory of health and functional outcomes in children following a critical illness, define poor functional recovery, and evaluate predictors of poor recovery.

The Research Questions for this study are: 1) What are the health and functional outcomes in children affected by a critical illness, at 3 and 6 months following Pediatric Intensive Care Unit (PICU) discharge? 2) What defines poor functional recovery? 3) What are predictors of poor functional recovery in critically ill children? 4) What are the most important and relevant outcomes in critically ill children, from the patient and caregiver's point of view?

Study Design: Prospective Observational Mixed Methods Longitudinal Cohort Study Study Setting: Two Academic Pediatric Centres in Canada - McMaster Children's Hospital and London Health Sciences Centre.

ELIGIBILITY:
Inclusion Criteria:

* Age over 12 months to 17 years
* Admitted to PICU for at least 48 hours
* ≥ one organ dysfunction on admission
* Informed consent of patient/substitute decision maker, and patient assent were appropriate

Exclusion Criteria:

* Patients transferred directly from a neonatal intensive care unit prior to discharge home
* Patients who are already mobilizing well, or are at baseline functional status at time of screening
* Previous enrolment into this study
* Language barrier (i.e. no access to translation services)

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In order to enrol children at potential risk for the outcomes of interest, and avoid "healthier" participants with short PICU stays, we considered the following: the patient should have: a) a minimum age (when one is expected to be ambulatory/mobilizing), and b) a threshold severity of illness. In order to understand how different subsets of PICU populations are affected by critical illness, we chose not to restrict the selection of patients to a specific diagnosis, nor did we exclude patients with underlying functional or cognitive abnormalities at baseline. This study will evaluate the epidemiology of recovery in a general critically ill pediatric population over time.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Functional Recovery | In the first 6 months following Pediatric Intensive Care Unit Discharge
  Functional Status will be measured at PICU discharge, 3 and 6 months post discharge using the following measurement tools: Pediatric Evaluation of Disability Inventory (PEDI), and the Participation and Environment Measure - children and youth versions (PEM-CY/YC-PEM).
Predictors of Functional Recovery | 6 months post PICU discharge
  The following hypothesized determinants of functional recovery will be evaluated: age, critical illness severity, pre-admission co-morbid status, PICU discharge functional status, and time to rehabilitation.

SECONDARY OUTCOMES:
Additional components of functional health | The first 6 months post PICU discharge
  Functional Health Status will be measured using the International Classification of Functioning, Disability and Health (ICF) framework (www.who.int/icidh/). In addition to the primary outcome measurements, the following will be assessed: Caregiver burden using the Pediatric Inventory for Parents; and Health Related Quality of Life using KIDSCREEN. The following secondary outcomes of interest will also be measured: Short-term PICU outcomes (i.e. duration of ventilation, length of stay, severity of organ dysfunction, morbidities attributable to delayed mobilization); mortality, health care utilization, and Pediatric Cerebral performance category and Pediatric Overall Performance scores in the 6 months post PICU discharge.

OTHER OUTCOMES:
Audit of Patient Centeredness of Outcomes | 6 months post PICU discharge
  Qualitative methodology will be used in this study to understand what is important to patients and families following survival from a critical illness, and if our selected outcomes of interest for this study are aligned with what patients and families consider meaningful and important. Patient and caregiver interviews will be conducted for this purpose in the 6 months following PICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MB, BCh, MSc, Principal Investigator — McMaster University; Canadian Critical Care Trials Group
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Sciences, London, Ontario

REFERENCES:
- [Derived] Jarvis JM, Fayed N, Fink EL, Choong K, Khetani MA. Caregiver dissatisfaction with their child's participation in home activities after pediatric critical illness. BMC Pediatr. 2020 Sep 2;20(1):415. doi: 10.1186/s12887-020-02306-3. PMID 32878614
- [Derived] Jarvis JM, Gurga AR, Lim H, Cameron J, Gorter JW, Choong K, Khetani MA. Caregiver Strategy Use to Promote Children's Home Participation After Pediatric Critical Illness. Arch Phys Med Rehabil. 2019 Nov;100(11):2144-2150. doi: 10.1016/j.apmr.2019.05.034. Epub 2019 Jul 3. PMID 31278925
- [Derived] Jarvis JM, Choong K, Khetani MA. Associations of Participation-Focused Strategies and Rehabilitation Service Use With Caregiver Stress After Pediatric Critical Illness. Arch Phys Med Rehabil. 2019 Apr;100(4):703-710. doi: 10.1016/j.apmr.2018.11.017. Epub 2018 Dec 19. PMID 30578773
- [Derived] Khetani MA, Albrecht EC, Jarvis JM, Pogorzelski D, Cheng E, Choong K. Determinants of change in home participation among critically ill children. Dev Med Child Neurol. 2018 Aug;60(8):793-800. doi: 10.1111/dmcn.13731. Epub 2018 Mar 25. PMID 29574916